CLINICAL TRIAL: NCT07343245
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetics Drug-Drug Interaction of DW4421 and 3 NSAIDs in Healthy Adult Volunteers
Brief Title: A Phase 1 Clinical Trial to Evaluate the Safety and DDI of DW4421 and 3 NSAIDs
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DW4421-102
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1, A (Experimental)
  Interventions: Drug: DW4421; Drug: DW4421-N1
- Cohort 1, B (Experimental)
  Interventions: Drug: DW4421; Drug: DW4421-N1
- Cohort 2, C (Experimental)
  Interventions: Drug: DW4421; Drug: DW4421-N2
- Cohort 2, D (Experimental)
  Interventions: Drug: DW4421; Drug: DW4421-N2
- Cohort 3, E (Experimental)
  Interventions: Drug: DW4421; Drug: DW4421-N3
- Cohort 3, F (Experimental)
  Interventions: Drug: DW4421; Drug: DW4421-N3

INTERVENTIONS:
Drug: DW4421 — QD
Drug: DW4421-N1 — BID
  Arms: Cohort 1, A; Cohort 1, B
Drug: DW4421-N2 — BID
  Arms: Cohort 2, C; Cohort 2, D
Drug: DW4421-N3 — QD
  Arms: Cohort 3, E; Cohort 3, F

SUMMARY:
Drug-Drug Interaction between DW4421 and three different kinds of NSAIDs

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 19 to 50 (inclusive) years, at the time of screening.
* Subjects weighing between 50 kg and 90 kg with BMI between 18 and 27 kg/m2 (inclusive) at screening visit.

Exclusion Criteria:

* Those who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss | Baseline to Day 13 or Day 15
AUCτ,ss | Baseline to Day 13 or Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea